CLINICAL TRIAL: NCT03429556
Title: A Phase 2 Study to Evaluate Safety and Efficacy of EB-001 Intramuscular (IM) Injections in Reducing Musculoskeletal Pain in Subjects Undergoing Elective Abdominoplasty Surgery
Brief Title: Study to Evaluate Botulinum Neurotoxin Serotype E (EB-001) in Reducing Musculoskeletal Pain in Abdominoplasty
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Sponsor decision to terminate early
Sponsor: Allergan (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: EB001-ABD201
Record Dates: First submitted 2018-02-06; First posted 2018-02-12 (Actual); Results first posted 2019-08-05 (Actual); Last update posted 2019-08-05 (Actual); Status verified 2019-08

CONDITIONS: Abdominoplasty
Keywords: pain, neurotoxin
MeSH Terms: conditions — Pain

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Placebo (Placebo Comparator): Placebo (sterile saline solution 0.9% Sodium Chloride Injection) injected into RA muscles during abdominoplasty surgery.
  Interventions: Drug: Placebo
- Botulinum Neurotoxin Serotype E Dose 1 (Experimental): Single botulinum neurotoxin serotype E Dose 1 injection into RA muscles during abdominoplasty surgery.
  Interventions: Biological: Botulinum Neurotoxin Serotype E
- Botulinum Neurotoxin Serotype E Dose 2 (Experimental): Single botulinum neurotoxin serotype E Dose 2 injection into RA muscles during abdominoplasty surgery.
  Interventions: Biological: Botulinum Neurotoxin Serotype E
- Botulinum Neurotoxin Serotype E Dose 3 (Experimental): Single botulinum neurotoxin serotype E Dose 3 injection into RA muscles during abdominoplasty surgery.
  Interventions: Biological: Botulinum Neurotoxin Serotype E

INTERVENTIONS:
Biological: Botulinum Neurotoxin Serotype E — Single botulinum neurotoxin serotype E injection into RA muscles during abdominoplasty surgery.
  Other Names: EB-001; BoNT/E
  Arms: Botulinum Neurotoxin Serotype E Dose 1; Botulinum Neurotoxin Serotype E Dose 2; Botulinum Neurotoxin Serotype E Dose 3
Drug: Placebo — Placebo (sterile saline solution 0.9% Sodium Chloride Injection) injected into RA muscles during abdominoplasty surgery.
  Arms: Placebo

SUMMARY:
To determine the safety and efficacy of single intra-operative treatment of Botulinum Neurotoxin Serotype E (EB-001) intramuscular (IM) injections into the Rectus Abdominus (RA) in participants undergoing abdominoplasty.

ELIGIBILITY:
Inclusion Criteria:

1. Men or women 23 to 55 years of age, inclusive
2. Scheduled to undergo elective abdominoplasty surgery with full length plication from xyphoid to pubis, and removal of skin/fat flap under general anesthesia (endotracheal or otherwise) without liposuction
3. American Society of Anesthesiologist (ASA) Physical Class 1-2.

Exclusion Criteria:

1. History of prior major abdominal surgery as judged by the investigator
2. Pre-existing lung disease that could impact participant safety in the opinion of the investigator
3. Pre-existing disorders of the neuromuscular junction (myasthenia gravis, Eaton- Lambert syndrome, or amyotrophic lateral Sclerosis)
4. At high risk of deep vein thrombosis as judged by the investigators determined by a Caprini score of 3 or higher
5. Slow vital capacity that is below 80% of normal value for respective race, age, height, and gender or below 2.5 Liters (L) of absolute volume
6. Pulse oximetry below 95%
7. Body weight less than 50 kg (110 pounds) or a Body Mass Index (BMI) of ≥ 32
8. Reported use of any botulinum toxin within 3 months prior to the date of surgery
9. Use of long acting opioids within 3 days or any opioid medication within 24 hours prior to surgery
10. Aminoglycoside intake within 48 hours prior to or during surgery
11. Participants on anti-depressant or anti-psychotic medications
12. Reported pain score of 2 or more at screening on the 11-point scale numerical pain rating scale-administered after an activity (NPRS-A) following an activity after and walking approximately 10 feet.

Ages: 23 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 23 (Actual)
Dates: Start 2018-05-08 (Actual); Primary Completion 2018-07-10 (Actual); Study Completion 2018-07-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Joan-En Lin, Study Director — Allergan
Locations (2):
- United States (2):
  - Huntington Ambulatory Surgery Center, Pasadena, California
  - Lotus Clinical Research, LLC, Pasadena, California

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo: Placebo (sterile saline solution 0.9% Sodium Chloride Injection) injected into rectus abdominus (RA) muscles during abdominoplasty surgery.
Period: Overall Study
Arm/Group | Placebo | Botulinum Neurotoxin Serotype E Dose 1 | Botulinum Neurotoxin Serotype E Dose 2 | Botulinum Neurotoxin Serotype E Dose 3
Started | 12 | 4 | 4 | 3
Completed | 12 | 3 | 4 | 3
Not Completed | 0 | 1 | 0 | 0
Not completed — Lost to Follow-up | 0 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Safety Population included all participants exposed to any amount of study drug.
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Botulinum Neurotoxin Serotype E Dose 1 | Botulinum Neurotoxin Serotype E Dose 2 | Botulinum Neurotoxin Serotype E Dose 3 | Total
Number analyzed (Participants) | 12 | 4 | 4 | 3 | 23
Age, Continuous [Mean (Standard Deviation); unit: years] | 36.5 (5.2) | 33.0 (6.38) | 36.3 (7.72) | 41.0 (14.0) | 36.7 (3.29)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 4 | 4 | 3 | 22
  Male | 1 | 0 | 0 | 0 | 1
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 0 | 0 | 1 | 0 | 1
  Black or African American | 5 | 3 | 1 | 2 | 11
  White or Caucasian | 6 | 1 | 2 | 1 | 10
  Other/Mixed | 1 | 0 | 0 | 0 | 1
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Hispanic or Latino | 6 | 1 | 2 | 1 | 10
  Not Hispanic or Latino | 6 | 3 | 2 | 2 | 13

OUTCOME MEASURES:

1. Primary Outcome: Area Under the Curve (AUC) of Participant's Assessment of Pain Using the Numerical Pain Rating Scale (NPRS) at Rest Between 12 and 96 Hours Postsurgery (AUC12-96)
Description: The participant assessed their current pain using the 11-point NPRS where: 0=no pain to 10=worst pain imaginable. AUC was calculated using the standard trapezoidal rule.
Time Frame: Every 2 hours from 12 to 96 hours postsurgery
Population: Modified Intent-to-treat (mITT) population included all randomized and treated participants with at least one post-injection pain score.
Measure: Mean (Standard Deviation); unit: hour (hr)*score on a scale
Arm/Group | Placebo | Botulinum Neurotoxin Serotype E Dose 1 | Botulinum Neurotoxin Serotype E Dose 2 | Botulinum Neurotoxin Serotype E Dose 3
Number analyzed (Participants) | 11 | 1 | 4 | 3
hour (hr)*score on a scale | 321.18 (217.993) | 209.30 (NA) — Standard deviation (SD) was not calculated for 1 participant. | 415.40 (124.101) | 372.53 (135.799)

2. Secondary Outcome: AUC of Participant's Assessment of Pain Using the NPRS at Rest Between 0 and 96 Hours Postsurgery
Description: as for outcome 1
Time Frame: Every 2 hours from 0 to 96 hours postsurgery
Population: mITT population included all randomized and treated participants with at least one post-injection pain score.
Measure: Mean (Standard Deviation); unit: hr*score on a scale
Arm/Group | Placebo | Botulinum Neurotoxin Serotype E Dose 1 | Botulinum Neurotoxin Serotype E Dose 2 | Botulinum Neurotoxin Serotype E Dose 3
Number analyzed (Participants) | 11 | 1 | 4 | 3
hr*score on a scale | 403.80 (229.152) | 282.50 (NA) — SD was not calculated for 1 participant. | 506.83 (130.598) | 450.97 (139.769)

3. Secondary Outcome: AUC of Participant's Assessment of Pain Using the NPRS at Rest Between 0 and 72 Hours Postsurgery (AUC0-72)
Description: as for outcome 1
Time Frame: Every 2 hours from 0 to 72 hours postsurgery
Population: mITT population included all randomized and treated participants with at least one post-injection pain score.
Measure: Mean (Standard Deviation); unit: hr*score on a scale
Arm/Group | Placebo | Botulinum Neurotoxin Serotype E Dose 1 | Botulinum Neurotoxin Serotype E Dose 2 | Botulinum Neurotoxin Serotype E Dose 3
Number analyzed (Participants) | 11 | 1 | 4 | 3
hr*score on a scale | 338.91 (173.785) | 280.50 (NA) — SD was not calculated for 1 participant. | 416.70 (97.464) | 372.47 (86.226)

4. Secondary Outcome: AUC of Participant's Assessment of Pain Using the NPRS at Rest Between 0 and 48 Hours Postsurgery (AUC0-48)
Description: as for outcome 1
Time Frame: Every 2 hours from 0 to 48 hours postsurgery
Population: mITT population included all randomized and treated participants with at least one post-injection pain score.
Measure: Mean (Standard Deviation); unit: hr*score on a scale
Arm/Group | Placebo | Botulinum Neurotoxin Serotype E Dose 1 | Botulinum Neurotoxin Serotype E Dose 2 | Botulinum Neurotoxin Serotype E Dose 3
Number analyzed (Participants) | 11 | 1 | 4 | 3
hr*score on a scale | 253.53 (106.862) | 240.80 (NA) — SD was not calculated for 1 participant. | 283.20 (60.450) | 274.47 (32.686)

5. Secondary Outcome: AUC of Participant's Assessment of Pain Using the NPRS at Rest Between 0 and 24 Hours Postsurgery (AUC0-24)
Description: as for outcome 1
Time Frame: Every 2 hours from 0 to 24 hours postsurgery
Population: mITT population included all randomized and treated participants with at least one post-injection pain score.
Measure: Mean (Standard Deviation); unit: hr*score on a scale
Arm/Group | Placebo | Botulinum Neurotoxin Serotype E Dose 1 | Botulinum Neurotoxin Serotype E Dose 2 | Botulinum Neurotoxin Serotype E Dose 3
Number analyzed (Participants) | 11 | 1 | 4 | 3
hr*score on a scale | 144.49 (46.693) | 149.80 (NA) — The SD was not calculated due to less number of participants with data. | 155.53 (28.726) | 146.30 (21.717)

6. Secondary Outcome: AUC of Participant's Assessment of Pain Using the NPRS at Rest Between 12 and 24 Hours Postsurgery (AUC12-24)
Description: as for outcome 1
Time Frame: Every 2 hours from 12 to 24 hours postsurgery
Population: mITT population included all randomized and treated participants with at least one post-injection pain score.
Measure: Mean (Standard Deviation); unit: hr*score on a scale
Arm/Group | Placebo | Botulinum Neurotoxin Serotype E Dose 1 | Botulinum Neurotoxin Serotype E Dose 2 | Botulinum Neurotoxin Serotype E Dose 3
Number analyzed (Participants) | 11 | 1 | 4 | 3
hr*score on a scale | 61.91 (32.210) | 76.60 (NA) — SD was not calculated for 1 participant. | 64.10 (22.825) | 67.83 (18.827)

7. Secondary Outcome: Participants Overall Assessment of Pain Using the NPRS After Discharge
Description: The participant assessed their pain after discharge using the 11-point NPRS where: 0=no pain to 10=worst pain imaginable.
Time Frame: Days 6, 7, 8, 9, 10, 11, 12, 13, 14, 16, 18, 20, 22, 24 and 26
Population: mITT population included all randomized and treated participants with at least one post-injection pain score.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Placebo | Botulinum Neurotoxin Serotype E Dose 1 | Botulinum Neurotoxin Serotype E Dose 2 | Botulinum Neurotoxin Serotype E Dose 3
Number analyzed (Participants) | 11 | 1 | 4 | 3
score on a scale
  Day 6 | 2.3 (1.66) | 0.0 (NA) — SD was not calculated for 1 participant. | 6.0 (1.83) | 2.3 (2.08)
  Day 7 | 2.3 (2.78) | 0.0 (NA) — SD was not calculated for 1 participant. | 3.8 (0.50) | 3.0 (3.00)
  Day 8 | 1.8 (1.79) | 0.0 (NA) — SD was not calculated for 1 participant. | 3.5 (1.73) | 3.0 (3.00)
  Day 9 | 2.1 (2.62) | 0.0 (NA) — SD was not calculated for 1 participant. | 5.3 (1.50) | 1.5 (2.12)
  Day 10 | 1.8 (1.92) | 0.0 (NA) — SD was not calculated for 1 participant. | 4.0 (0.82) | 1.5 (2.12)
  Day 11 | 1.8 (2.28) | 0.0 (NA) — SD was not calculated for 1 participant. | 3.3 (1.50) | 1.5 (2.12)
  Day 12 | 1.7 (1.87) | 0.0 (NA) — SD was not calculated for 1 participant. | 2.5 (1.29) | 1.5 (2.12)
  Day 13 | 1.7 (1.73) | 0.0 (NA) — SD was not calculated for 1 participant. | 3.0 (0.00) | 2.0 (2.83)
  Day 14 | 1.7 (1.94) | 0.0 (NA) — SD was not calculated for 1 participant. | 2.3 (1.71) | 2.0 (2.83)
  Day 16 | 1.9 (2.47) | 0.0 (NA) — SD was not calculated for 1 participant. | 2.0 (0.82) | 1.5 (2.12)
  Day 18 | 1.6 (2.26) | 0.0 (NA) — SD was not calculated for 1 participant. | 1.8 (0.96) | 1.5 (2.12)
  Day 20 | 1.6 (2.20) | 0.0 (NA) — SD was not calculated for 1 participant. | 1.8 (0.96) | 1.5 (2.12)
  Day 22 | 1.1 (1.73) | 0.0 (NA) — SD was not calculated for 1 participant. | 1.0 (1.41) | 1.5 (2.12)
  Day 24 | 1.5 (2.45) | 0.0 (NA) — SD was not calculated for 1 participant. | 1.0 (1.41) | 2.0 (2.83)
  Day 26 | 1.3 (1.98) | 0.0 (NA) — SD was not calculated for 1 participant. | 1.0 (1.41) | 1.5 (2.12)

8. Secondary Outcome: Participant's Overall Assessment of Pain Using the NPRS-Activity (NPRS-A)
Description: The participant assessed their pain using the 11-point NPRS-A, after sitting up in the bed unassisted at an angle of approximately ≥ 45 degrees, swinging legs out, putting feet down, standing up, and walking approximately 10 feet, where: 0=no pain to 10=worst pain imaginable.
Time Frame: 8, 16, 24, 30, 36, 42, 48, 54, 60, 66, 72.78.84, and 96 hours after surgery; Days 8, 15 and 29 after discharge
Population: mITT population included all randomized and treated participants with at least one post-injection pain score. Participants analyzed is the number of participants with data available for analysis at the given time point.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Placebo | Botulinum Neurotoxin Serotype E Dose 1 | Botulinum Neurotoxin Serotype E Dose 2 | Botulinum Neurotoxin Serotype E Dose 3
Number analyzed (Participants) | 11 | 1 | 4 | 3
score on a scale
  8 hours after surgery | 6.9 (2.74) | 5.0 (NA) — SD was not calculated for 1 participant. | 6.0 (2.45) | 6.3 (0.58)
  16 hours after surgery: number analyzed (Participants) | 11 | 1 | 0 | 1
  16 hours after surgery | 8.7 (1.53) | 4.0 (NA) — SD was not calculated for 1 participant. |  | 7.0 (NA) — SD was not calculated for 1 participant.
  24 hours after surgery | 6.6 (2.40) | 5.0 (NA) — SD was not calculated for 1 participant. | 7.5 (1.29) | 6.3 (0.58)
  30 hours after surgery | 6.5 (2.45) | 5.0 (NA) — SD was not calculated for 1 participant. | 7.0 (2.16) | 5.0 (2.00)
  36 hours after surgery | 6.3 (1.89) | 4.0 (NA) — SD was not calculated for 1 participant. | 6.5 (1.29) | 6.3 (0.58)
  42 hours after surgery: number analyzed (Participants) | 11 | 0 | 0 | 0
  42 hours after surgery | 5.8 (1.47) |  |  |
  48 hours after surgery | 4.3 (1.50) | 3.0 (NA) — SD was not calculated for 1 participant. | 5.3 (1.71) | 3.7 (1.53)
  54 hours after surgery | 4.8 (1.20) | 2.0 (NA) — SD was not calculated for 1 participant. | 6.3 (3.10) | 4.0 (2.00)
  60 hours after surgery | 6.3 (2.75) | 3.0 (NA) — SD was not calculated for 1 participant. | 6.0 (1.41) | 3.3 (2.52)
  66 hours after surgery: number analyzed (Participants) | 11 | 0 | 0 | 0
  66 hours after surgery | 4.7 (3.20) |  |  |
  72 hours after surgery | 3.7 (2.45) | 0.0 (NA) — SD was not calculated for 1 participant. | 4.0 (2.71) | 3.0 (1.73)
  78 hours after surgery | 3.6 (2.62) | 0.0 (NA) — SD was not calculated for 1 participant. | 4.5 (2.08) | 3.3 (2.08)
  84 hours after surgery | 4.5 (3.32) | 1.0 (NA) — SD was not calculated for 1 participant. | 5.0 (1.15) | 3.0 (2.65)
  96 hours after surgery | 2.4 (1.81) | 0.0 (NA) — SD was not calculated for 1 participant. | 3.5 (1.29) | 3.3 (3.06)
  Day 8 after discharge | 2.1 (2.20) | 1.0 (NA) — SD was not calculated for 1 participant. | 4.8 (1.71) | 3.3 (3.06)
  Day 15 after discharge | 1.6 (1.77) | 0.0 (NA) — SD was not calculated for 1 participant. | 3.8 (2.99) | 2.7 (2.31)
  Day 29 after discharge: number analyzed (Participants) | 11 | 0 | 4 | 1
  Day 29 after discharge | 1.5 (1.97) |  | 0.5 (0.58) | 0.0 (NA) — SD was not calculated for 1 participant.

9. Secondary Outcome: Number of Participants by Patient Global Assessment (PGA) of Pain Control Score Categories
Description: The participant assessed their overall pain control in the past 24 hours using the PGA 4-point scale where: 0=poor, 1=fair, 2=good and 3=excellent.
Time Frame: Days 5, 8, 15 and 29
Population: mITT population included all randomized and treated participants with at least one post-injection pain score.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Botulinum Neurotoxin Serotype E Dose 1 | Botulinum Neurotoxin Serotype E Dose 2 | Botulinum Neurotoxin Serotype E Dose 3
Number analyzed (Participants) | 11 | 1 | 4 | 3
Participants
  Day 5: PGA score 3 | 7 | 1 | 2 | 1
  Day 5: PGA score 2 | 4 | 0 | 2 | 1
  Day 5: PGA score 1 | 0 | 0 | 0 | 1
  Day 5: PGA score 0 | 0 | 0 | 0 | 0
  Day 8: PGA score 3 | 7 | 1 | 0 | 1
  Day 8: PGA score 2 | 4 | 0 | 2 | 0
  Day 8: PGA score 1 | 0 | 0 | 1 | 2
  Day 8: PGA score 0 | 0 | 0 | 1 | 0
  Day 15: PGA score 3 | 8 | 1 | 2 | 1
  Day 15: PGA score 2 | 3 | 0 | 1 | 1
  Day 15: PGA score 1 | 0 | 0 | 1 | 1
  Day 15: PGA score 0 | 0 | 0 | 0 | 0
  Day 29: PGA score 3 | 9 | 1 | 3 | 1
  Day 29: PGA score 2 | 2 | 0 | 1 | 2
  Day 29: PGA score 1 | 0 | 0 | 0 | 0
  Day 29: PGA score 0 | 0 | 0 | 0 | 0

10. Secondary Outcome: Number of Doses of Rescue Medications Used
Time Frame: Up to 96 hours postsurgery
Population: mITT population included all randomized and treated participants with at least one post-injection pain score.
Measure: Mean (Standard Deviation); unit: doses
Arm/Group | Placebo | Botulinum Neurotoxin Serotype E Dose 1 | Botulinum Neurotoxin Serotype E Dose 2 | Botulinum Neurotoxin Serotype E Dose 3
Number analyzed (Participants) | 11 | 1 | 4 | 3
doses
  Oxycodone | 9.7 (5.92) | 5.0 (NA) — SD was not calculated for 1 participant. | 11.8 (5.68) | 11.7 (4.93)
  Opioid | 14.2 (7.40) | 8.0 (NA) — SD was not calculated for 1 participant. | 15.8 (6.90) | 16.0 (6.08)

ADVERSE EVENTS:
Time Frame: Up to 31 days
Description: Safety Population included all participants exposed to any amount of study drug.
Arm/Group | Placebo | Botulinum Neurotoxin Serotype E Dose 1 | Botulinum Neurotoxin Serotype E Dose 2 | Botulinum Neurotoxin Serotype E Dose 3
All-Cause Mortality (participants affected / at risk) | 0/12 | 0/4 | 0/4 | 0/3
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/4 | 0/4 | 0/3
Other Adverse Events (participants affected / at risk) | 8/12 | 3/4 | 4/4 | 3/3
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=12) | Botulinum Neurotoxin Serotype E Dose 1 (N=4) | Botulinum Neurotoxin Serotype E Dose 2 (N=4) | Botulinum Neurotoxin Serotype E Dose 3 (N=3)
Nausea (Gastrointestinal disorders) | 6 | 1 | 2 | 2
Constipation (Gastrointestinal disorders) | 2 | 1 | 2 | 0
Vomiting (Gastrointestinal disorders) | 1 | 1 | 1 | 0
Dyspepsia (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 1 | 1 | 0
Pruritus generalised (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 2 | 0 | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 2 | 0
Headache (Nervous system disorders) | 5 | 1 | 1 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 2
Seroma (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Transaminases increased (Investigations) | 0 | 1 | 0 | 0
Depressed mood (Psychiatric disorders) | 0 | 1 | 0 | 0
Vaginal haemorrhage (Reproductive system and breast disorders) | 0 | 0 | 1 | 0
Food allergy (Immune system disorders) | 1 | 0 | 0 | 0
Tooth infection (Infections and infestations) | 1 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
A disclosure restriction on the PI is that the sponsor can review results communications prior to public release and can embargo communications regarding trial results for a period that is less than or equal to 90 days from the time submitted to the sponsor for review. The sponsor cannot require changes to the communication and cannot extend the embargo.

DOCUMENTS (2):
  • Study Protocol (2018-09-28): https://cdn.clinicaltrials.gov/large-docs/56/NCT03429556/Prot_000.pdf
  • Statistical Analysis Plan (2018-05-09): https://cdn.clinicaltrials.gov/large-docs/56/NCT03429556/SAP_001.pdf